CLINICAL TRIAL: NCT05686317
Title: A Randomized, Sham-controlled Clinical Trial for Evaluation of the Edwards APTURE Transcatheter Shunt System (ALT-FLOW II)
Brief Title: ALT-FLOW II Trial of the Edwards APTURE Transcatheter Shunt System
Acronym: ALT-FLOW II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-06
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- APTURE shunt + medical therapy (Experimental)
  Interventions: Device: Edwards APTURE transcatheter shunt system
- Sham + medical therapy (Sham Comparator)
  Interventions: Diagnostic Test: Sham procedure

INTERVENTIONS:
Device: Edwards APTURE transcatheter shunt system — Treatment with APTURE shunt
  Arms: APTURE shunt + medical therapy
Diagnostic Test: Sham procedure — CS angiography
  Arms: Sham + medical therapy

SUMMARY:
This is a prospective, multi-center, randomized, sham-controlled, double-blinded (participant and outcomes assessor) clinical trial.

DETAILED DESCRIPTION:
The objectives of this trial are to assess the safety, performance, and effectiveness of the Edwards APTURE transcatheter shunt system when used for the treatment of patients with heart failure with preserved (HFpEF) or mildly reduced (HFmrEF) ejection fraction (LVEF >40%) who remain symptomatic despite guideline-directed medical therapy (GDMT)

ELIGIBILITY:
Key Inclusion Criteria:

• Symptomatic heart failure

1. A primary diagnosis of HFmrEF or HFpEF (LVEF > 40%), and
2. NYHA class II to ambulatory NYHA class IV (IVa), and
3. Documentation of at least one of the following from the date of initial informed consent or date of enrollment:

i. Within the prior 12 months, EITHER:

* HF hospital admission (with HF as the primary or secondary diagnosis)
* Treatment with intravenous (IV) or intensification of oral diuretics for HF

ii. Within the prior 6 months, EITHER:

* BNP value > 35 pg/ml in normal sinus rhythm (NSR) or paroxysmal atrial fibrillation (AF)
* BNP > 125 pg/ml for permanent or long-term persistent AF
* NT-proBNP > 125 pg/ml in NSR or paroxysmal AF
* NT-proBNP > 375 pg/ml for permanent or long-term persistent AF d. There is objective evidence of cardiogenic pulmonary congestion based on hemodynamic criteria obtained by right heart catheterization (RHC) at exercise, and confirmed by hemodynamics core lab as: As measured at end-expiration, pulmonary capillary wedge pressure (PCWP) at ≥ 20 Watts exercise (PCWP ≥ 20W) is elevated to ≥ 25 mmHg and exceeds [the corresponding] right atrial pressure (RAP) by ≥ 8 mmHg • In the judgment of the treating physician and the Central Screening Committee the patient is on GDMT for HFpEF/HFmrEF for >30 days prior to screening and baseline assessments, that is expected to be maintained without change for 6 months.

Key Exclusion Criteria:

* Severe heart failure defined as one or more of the below:

  1. ACC/AHA/ESC Stage D HF, non-ambulatory NYHA Class IV HF
  2. If Body Mass Index (BMI) < 30, cardiac index < 2.0 L/min/m2
  3. If BMI ≥ 30, cardiac index < 1.8 L/min/m2
  4. Inotropic infusion (continuous or intermittent) within the past 6 months
  5. Patient is on the cardiac transplant waiting list
  6. Prior diagnosis of HF with reduced ejection fraction (HFrEF), including patients with improvement in LVEF to > 40%
* Valve disease:

  1. Degenerative mitral regurgitation > moderate
  2. Functional or secondary mitral valve regurgitation defined as grade > moderate
  3. Mitral stenosis > mild
  4. Primary or secondary tricuspid valve regurgitation defined as grade > moderate
  5. Aortic valve disease defined as aortic regurgitation grade > moderate or aortic stenosis > moderate
* More than mild right ventricular (RV) dysfunction as determined by the echo core lab, taking into account the following available parameters:

  1. Tricuspid annular plane systolic excursion (TAPSE) <1.4 cm, or
  2. RV size ≥ LV size
  3. Right ventricular ejection fraction (RVEF) < 35%; or
  4. Imaging or clinical evidence of congestive hepatopathy
* Mean right atrial pressure (mRAP) > 15 mmHg at rest
* Pulmonary vascular resistance (PVR) ≥ 5.0 WU
* BMI ≥ 45
* Myocardial infarction (MI) and/or any therapeutic invasive, non-valvular cardiovascular procedure within past 3 months or current indication for coronary revascularization
* Stroke, transient ischemic attack (TIA), deep vein thrombosis (DVT) or pulmonary embolus within the past 6 months
* Renal insufficiency as determined by creatinine (sCr) level > 2.5 mg/dL or estimated glomerular filtration rate (eGFR) < 25ml/min/1.73 m2 by CKD-Epi equation; or currently requiring dialysis
* Performance of the six-minute walk test (6MWT) with a distance < 50m OR > 450m
* Active endocarditis or infection requiring intravenous antibiotics within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Device + Medical Therapy: Subjects with Early Major Adverse Events | 30 days
  Shunt implant safety: proportion of patients in the APTURE shunt group without any serious device or procedure-related (CEC adjudicated) complications (i.e., Major Adverse Cardiovascular, Cerebrovascular, and Renal Events [MACCRE]; at 30 days post index procedure or hospital discharge, whichever is later.
Mean change in PCWL from baseline at 6 months | 6-months
  Hemodynamic Effectiveness: change in pulmonary capillary wedge during load (PCWL, mmHg/W/kg) from baseline at 6 months.

SECONDARY OUTCOMES:
KCCQ-OSS change from baseline at 6-month follow-up | 6-months
  Change in Kansas City Cardiomyopathy Questionnaire - Overall Summary Score (KCCQ-OSS) from baseline at 6-month follow-up.
Proportion of individual patient success defined as being free from death, disabling stroke, and HF hospitalization with at least (≥) a 15-point improvement from baseline KCCQ-OSS or at least (≥) a 25m improvement from baseline 6MWT. | 6-months
6MWT change from baseline at 6-month follow-up | 6-months
  Chang in 6-Minute Walk Test (6MWT) from baseline at 6-month follow-up

CONTACTS AND LOCATIONS:
Locations (33):
- United States (23):
  - University of California Irvine, Irvine, California
  - University of California San Diego, La Jolla, California
  - Scripps Health, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Ascension Illinois Heart and Vascular Medical Group, Elk Grove, Illinois
  - Northwestern University, Evanston, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Buffalo, Buffalo, New York
  - St. Francis Hospital & Heart Center, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Christ Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Oregon Health and Science University, Oregon City, Oregon
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina Charleston, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - Benaroya Virginia Mason, Seattle, Washington
- Instituto do Coracao da Universidade de Sao Paulo, São Paulo, Brazil
- Canada (2):
  - The Ottawa Hospital, Ottawa, Canada
  - St. Michael's Hospital, Toronto, Canada
- Germany (5):
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen
  - Herzzentrum Universitätsklinikum Köln, Cologne
  - Herzzentrum Dresden GmbH Universitätsklinik für Innere Medizin und Kardiologie, Dresden
  - Universitätsklinikum Heidelberg Medizinische Klinik, Heidelberg
  - Johannes Gutenberg Universitaet Mainz, Mainz
- Switzerland (2):
  - Inselspital Bern, Bern, Switzerland
  - Universitätsspital Basel, Basel

IPD SHARING:
Plan to Share IPD: No